CLINICAL TRIAL: NCT06363630
Title: A Phase 1, Open-label, 2-part, 2-period, Fixed-sequence, Crossover Study to Evaluate the Effect of Cytochrome P450 (CYP) 3A Inhibitor (Itraconazole) and Inducer (Rifampin) on the Pharmacokinetics of Golcadomide (BMS-986369) in Healthy Participants
Brief Title: A Study to Evaluate the Effect of Cytochrome P450 (CYP) 3A Inhibitor (Itraconazole) and Inducer (Rifampin) on the Drug Levels of Golcadomide (BMS-986369) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA073-1000
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: pharmacokinetics; BMS-986369; CC-99282; healthy
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental)
  Interventions: Drug: Itraconazole; Drug: Golcadomide
- Part 2 (Experimental)
  Interventions: Drug: Rifampin; Drug: Golcadomide

INTERVENTIONS:
Drug: Itraconazole — Specified dose on specified days.
  Arms: Part 1
Drug: Rifampin — Specified dose on specified days
  Arms: Part 2
Drug: Golcadomide — Specified dose on specified days
  Other Names: BMS-986369

SUMMARY:
The purpose of this study is to evaluate the drug-drug interaction (DDI) potential of coadministration of itraconazole or rifampin on the single dose drug levels of golcadomide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female non smoking participants, of any race, as determined by the investigator to have no clinically significant deviation from normal, in medical history and physical examination which correspond to a condition that could potentially increase the risk for the participants, or jeopardize the integrity of the study data, in 12-lead ECG measurements, vital signs, and clinical laboratory determinations, at screening and at check-in.
* Body mass index (BMI) 18.0 to 33.0 kg/m2, inclusive. BMI = weight (kg)/(height [m])2 for participants.
* Participant is afebrile (febrile is defined as ≥ 38°C or ≥ 100.4°F), with systolic blood pressure ≥ 90 and ≤ 140 mmHg, diastolic blood pressure ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 90 beats per minute at screening, confirmed by repeat, as per clinical site's standard.
* Must have a normal or clinically acceptable 12-lead ECG at screening: Participants must have a corrected QT interval using QTcF value ≤ 450 msec.
* Absolute neutrophil counts must be greater than 2,500/μL at screening and Day -1.
* Must have adequate laboratory test results for renal and hepatic function as assessed by the PI (Principal Investigator). Laboratory testing may be repeated to find all possible well-qualified participants.

Exclusion Criteria:

* Any significant acute or chronic medical illness that presents a potential risk to the participant in the opinion of the investigator and/or may compromise the objectives of the study.
* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular (CV), peripheral vascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary (GU) abnormalities/diseases.
* Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME). Appendectomy and cholecystectomy are acceptable. Prior procedures of unclear ADME significance should be reviewed with the Sponsor's Medical Monitor.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to Day 67
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to Day 67
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 67

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 69
Number of participants with physical exam abnormalities | Up to Day 69
Number of participants with vital sign abnormalities | Up to Day 69
Number of participants with clinical laboratory safety test abnormalities | Up to Day 69
Number of participants with electrocardiogram abnormalities | Up to Day 69
Number of participants with concomitant medications | Up to Day 69
Number of participants with concomitant procedures | Up to Day 69
Time of maximum observed plasma concentration (Tmax) | Up to Day 67
Apparent terminal phase half-life (T-HALF) | Up to Day 67
Apparent total body clearance (CLT/F) | Up to Day 67
Apparent volume of distribution (Vz/F) | Up to Day 67

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0002, Atlanta, Georgia
  - Local Institution - 0001, Lenexa, Kansas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com